CLINICAL TRIAL: NCT02301169
Title: A Study to Investigate the Effects of T4P1001 Treatment in Patients With Peripheral Neuropathic Pain
Brief Title: A Study to Investigate the Effects of a New Treatment in Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tools4Patient (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: T1001-01
Record Dates: First submitted 2014-11-14; First posted 2014-11-25 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Peripheral Neuropathies
Keywords: Pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T4P1001 (Active Comparator)
  Interventions: Behavioral: Heat pain stimuli A; Behavioral: Video A; Drug: Administration of T4P1001 capsules
- Placebo (Sham Comparator)
  Interventions: Behavioral: Heat pain stimuli B; Behavioral: Video B; Drug: Administration of placebo capsules

INTERVENTIONS:
Behavioral: Heat pain stimuli A
  Arms: T4P1001
Behavioral: Video A
  Arms: T4P1001
Drug: Administration of T4P1001 capsules — This treatment is given as add on therapy to patients' regular analgesic
  Arms: T4P1001
Behavioral: Heat pain stimuli B
  Arms: Placebo
Behavioral: Video B
  Arms: Placebo
Drug: Administration of placebo capsules — This treatment is given as add on therapy to patients' regular analgesic
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial conducted in patients suffering from chronic pain is to study the relationship between individual patients' profile and their analgesic response.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of at least 18 years of age
* Body weight of more than 40 kg and less than 120 kg with a BMI between 19-31 kg/m2 inclusive
* Diagnosed with Peripheral Neuropathic Pain (PNP) since at least 6 months
* Being affiliated with the national welfare system
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by the relevant Ethics Committee (EC) governing the study site

PNP disease diagnosis inclusion criteria:

* Patient with chronic PNP supported by a distinct neuroanatomical plausible distribution with sensory signs and symptoms, and consecutive to one of the following causes: a traumatic event, a surgical procedure (excluding limb amputation), radiculopathy, post-herpetic or post-zooster neuralgia, diabetic polyneuropathy or post-anticancer chemotherapy. Diagnosis will have to be confirmed by the DN4 questionnaire at the screening visit (pain is considered as neuropathic if DN4 score ≥ 4)
* Pain present since at least 6 months
* Patients will be required to have a score between 4 and 8 inclusive on the mean Average Pain Score (APS) Numeric Rating Scale (NRS) during the baseline period preceding randomization (data collected in patient diary) and to have completed at least 4 days of pain assessment

Exclusion Criteria:

* Pregnant, breastfeeding, or willing to be pregnant within 2 months
* With a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the patient's participation in the study
* Uncontrolled epilepsy
* Any current primary psychiatric condition, including major depression or major personality disorders (such as Axe II of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV); personality disorders and mental retardation)
* Alcohol dependence or regular use of known drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and phencyclidine)
* Acute disease state within 7 days before Visit 2
* Any other relevant medical disorder likely to interfere with the trial or represent a risk for the patient
* Any close relationship with the Investigators or the Sponsor (i.e. belonging to immediate family or subordination link)
* Patient under legal protection, according to the national law
* Patient currently enrolled in a clinical trial involving use of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study, or in an exclusion period according to national law

Exclusion criteria related to PNP:

* Neuropathic pain due to trigeminal neuralgia, central pain, complex regional pain syndrome and phantom limb pain
* Plan to have a session of physiotherapy or comportemental therapy such as gestion of pain, hypnosis, sophrology, meditation program during the study
* Have initiated or have planned an electrical stimulation (or neurostimulation) therapy within 2 weeks prior to Visit 1 or during the study period up to Visit 5
* Patient changed his/her " regular therapy " in the last 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pereira, Study Director — Tools4Patient
Locations (1):
- CIC Clermont-Ferrand, CHU Clermont-Ferrand, Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Groups:
- T4P1001: Heat pain stimuli A
  Video A
  Administration of T4P1001 capsules: This treatment is given as add on therapy to patients' regular analgesic
- Placebo: Heat pain stimuli B
  Video B
  Administration of placebo capsules: This treatment is given as add on therapy to patients' regular analgesic
Period: Overall Study
Arm/Group | T4P1001 | Placebo
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T4P1001 | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.3) | 55.5 (12.7) | 56.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Patient 's Change From Baseline of Pain Severity as Measured by the Weekly Means of the Daily Average Pain Scores (APS) During 4 Weeks of Treatment
Description: 11-point Numeric Rating Scale (NRS). Scale from 0 to 10, 0 meaning no pain, 10 pain as bad as you can imagine. Lower values represent a better outcome. Unit: arithmetic average of 7 days of a 11-point NRS
Time Frame: Time zero equals baseline (Day 1) up to Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 20 | 21
units on a scale | 0.87 (1.49) | 0.5 (1.43)
Statistical Analysis 1: Comparison: T4P1001 vs Placebo; Test type: Non-Inferiority or Equivalence — Null hypothesis: no difference in mean change from baseline to day 42 of pain severity as measured by weekly means of the daily Average Pain Score (APS), T4P1001 compared with placebo; p = 0.4162, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment group comparisons; Welch two sample t-test; Mean Difference (Final Values) = 0.3748299, 95% CI 2-sided [-0.5479411 to 1.2976010]

2. Secondary Outcome: Patient 's Change From Baseline of Pain Severity as Measured by the Weekly Means of the Daily Worst Pain Scores (WPS)
Description: 11-point Numeric Rating Scale (NRS) Scale from 0 to 10, 0 meaning no pain, 10 pain as bad as you can imagine. Lower values represent a better outcome. Unit: arithmetic average of 7 days of a 11-point NRS
Time Frame: Time zero equals baseline (Day 1) up to Day 42
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 20 | 21
units on a scale | 0.78 (1.45) | 0.65 (1.53)
Statistical Analysis 1: Comparison: T4P1001 vs Placebo; Test type: Non-Inferiority or Equivalence — Null hypothesis: no difference in mean change from baseline to day 42 of pain severity as measured by weekly means of the daily Worst Pain Score (WPS), T4P1001 compared with placebo; p = 0.7887, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Welch two sample t-test; Mean Difference (Final Values) = 0.1255102, 95% CI 2-sided [-0.8152493 to 1.0662697]

3. Secondary Outcome: Patient's Change From Baseline of Investigator Global Assessment of Change (IGAC)
Description: IGAC is an investigator subjective evaluation of patient condition using a NRS from 0 to 10 with 0 meaning best and 10 worst Lower values represent a better outcome.
Time Frame: Time zero equals baseline (Day 1) up to Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 20 | 21
units on a scale | -0.15 (1.755) | -0.95 (2.459)
Statistical Analysis 1: Comparison: T4P1001 vs Placebo; Test type: Non-Inferiority or Equivalence — Null hypothesis: no difference in mean change from baseline to day 42 of pain severity as measured by Investigator Global Assessment of Change, T4P1001 compared with Placebo; p = 0.2353, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Welch two sample t-test; Mean Difference (Final Values) = 0.802381, 95% CI 2-sided [-0.5457743 to 2.1505362]

4. Secondary Outcome: Patient's Change of Pain Intensity After Heat Pain Stimuli From Baseline to End of Treatment Period
Description: 11-point Numeric Rating Scale (NRS) from 0 to 10; 0 meaning no pain, 10 pain as bad as you can imagine Lower values represent a better outcome Unit: arithmetic average on 6 reported scores per Visit.
Time Frame: Time zero equals baseline (Day 1) up to Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 20 | 21
units on a scale | 0.76 (1.003) | -0.01 (1.502)
Statistical Analysis 1: Comparison: T4P1001 vs Placebo; Test type: Non-Inferiority or Equivalence — Null hypothesis: no difference in mean change from baseline to day 42 of pain intensity measured after heat pain stimuli, T4P1001 compared with placebo; p = 0.06204, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Welch two sample t-test; Mean Difference (Final Values) = 0.7656429, 95% CI 2-sided [-0.0406744 to 1.5719601]

5. Secondary Outcome: Patient 's Change From Baseline of Pain Severity as Measured by the Weekly Means of the Brief Pain Inventory (BPI).
Description: Arithmetic average of 3 questions on an 11-point Numeric Rating Scale (NRS) from 0 to 10, 0 meaning no pain, 10 pain as bad as you can imagine.
  Lower values represent a better outcome
Time Frame: Time zero equals baseline (Day 1) up to Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | T4P1001 | Placebo
Number analyzed (Participants) | 20 | 21
units on a scale | 3.35 (5.422) | 1.67 (5.704)
Statistical Analysis 1: Comparison: T4P1001 vs Placebo; Test type: Non-Inferiority or Equivalence — Null hypothesis: no difference in mean change from baseline to day 42 of pain severity as measured by the Brief Pain Inventory (BPI), T4P1001 compared with placebo; p = 0.3386, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Welch two sample t-test; Mean Difference (Final Values) = 1.683333, 95% CI 2-sided [-1.831190 to 5.197857]

ADVERSE EVENTS:
Arm/Group | T4P1001 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 7/21 | 6/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T4P1001 (N=21) | Placebo (N=21)
Migraine (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 4 | 3
Cervical pain (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Specific agreement as part of Eureka project